CLINICAL TRIAL: NCT01731548
Title: Omitting Elective Nodal Irradiation and Irradiating Post-induction Versus Pre-induction Chemotherapy Tumor Extent for Limited-stage Small Cell Lung Cancer
Brief Title: A Prospective Randomized Study Comparing the Target Volume for Limited-stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-10-25
Record Dates: First submitted 2012-11-14; First posted 2012-11-21 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Carcinoma of Lung; Small Cell; Limited Stage
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study arm (Experimental): For patients who are randomized to study arm, (i.e. to irradiate the post-chemotherapy tumor extent) the clinical target volume-tumor (CTV-T) includes the post-chemotherapy gross tumor volume-tumor (GTV-T) with a margin of 0.8 cm.
  Chemotherapy includes etoposide 100mg/m2 d1-d3 combine with cisplatin 80mg/m2 d1 at 21-day interval for 4 cycles.
  Radiotherapy will be administered with cycle 3 chemotherapy（1.5 Gy twice daily to 45 Gy in 30 fractions over 3 weeks）
  Interventions: Radiation: hyperfractionated radiation therapy for both arms
- control arm (Active Comparator): For patients who are randomized to control arm, (i.e. to irradiate the pre-chemotherapy tumor extent) the clinical target volume-tumor (CTV-T) includes the pre-chemotherapy gross tumor volume-tumor (GTV-T) with a margin of 0.8 cm.
  Chemotherapy includes etoposide 100mg/m2 d1-d3 combine with cisplatin 80mg/m2 d1 at 21-day interval for 4 cycles.
  Radiotherapy will be administered with cycle 3 chemotherapy (1.5 Gy twice daily to 45 Gy in 30 fractions over 3 weeks).
  Interventions: Radiation: hyperfractionated radiation therapy for both arms

INTERVENTIONS:
Radiation: hyperfractionated radiation therapy for both arms — 1.5 Gy twice daily to 45 Gy in 30 fractions over 3 weeks for both arms

SUMMARY:
We hypothesized that the local control for both arms were not statistically significant, when irradiation to the post-induction chemotherapy tumor volume is compared with irradiation to the pre-induction chemotherapy tumor volume.While elective nodal irradiation will be omitted for both arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they had histologic or cytologic verification of small cell lung cancer (SCLC) and were radiographically confirmed limited-stage
* Patients with contralateral mediastinal and ipsilateral supraclavicular lymphadenopathy were also included.
* The patients should be between 18 and 75 years old without previous thoracic radiotherapy, chemotherapy or biotherapy.
* Karnofsky performance status was ≥ 80.
* Forced expiratory volume at 1 second (FEV1) ≥ 1 L.
* Had measurable or assessable disease.
* Neutrophilic granulocyte ≥ 1.5×109/L, haemoglobin ≥ 100 g/L, platelet count ≥ 100×109/L.
* Serum creatine and bilirubin < 1.5 × the upper normal limit (UNL), aminotransferase < 2 × UNL.
* Weight loss was less than 10% within 6 months before diagnosis.
* Written informed consent was required from all patients.

Exclusion Criteria:

* Patients were ineligible if they had a history of other malignant diseases except for non-melanomatous skin cancer and carcinoma in situ of the cervix, or any contraindications for chemoradiotherapy, malignant pleural and/or pericardial effusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2002-06; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
local-regional progression | at least 6 months

SECONDARY OUTCOMES:
overall survival | at least 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chen, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Sun Yat-Sen University, Cancer Center, Guangzhou, Guangdong, China